CLINICAL TRIAL: NCT01669304
Title: Pharmacologic Dissection of Vestibular Migraine and Chronic Subjective Dizziness: A Double-Blind Parallel Group Trial Comparing Response to Verapamil Versus Sertraline
Brief Title: Verapamil vs. Sertraline for Vestibular Migraine & Chronic Subjective Dizziness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey P. Staab, Associate Professor, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 12-002814
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Vestibular Migraine; Chronic Subjective Dizziness
Keywords: migraine variant; chronic dizziness; pharmacologic dissection
MeSH Terms: conditions — Migraine Disorders | interventions — Verapamil; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verapamil (Experimental): Verapamil extended release oral tablets administered in a flexible dose format ranging from 120 mg to 360 mg daily, as determined by severity of headache and dizziness.
  Interventions: Drug: Verapamil
- Sertraline (Experimental): Sertraline oral tablets administered in a flexible dose format ranging from 25 mg to 150 mg daily depending on severity of headache and dizziness.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Verapamil
  Other Names: Calan SR; Covera-HS; Isoptin SR; Verelan PM
  Arms: Verapamil
Drug: Sertraline
  Other Names: Zoloft
  Arms: Sertraline

SUMMARY:
Vestibular migraine (VM) and chronic subjective dizziness (CSD) commonly cause vertigo, unsteadiness and dizziness. Clinical investigators are studying these illnesses to understand them better. VM and CSD occur together in about 1/3 of patients. That makes it hard to diagnose them accurately and decide what treatments to use. As a result, doctors and patients may be confused about these diagnoses. The goal of this study was use two different medications to tease apart the symptoms of VM and CSD.

Patients who have VM and CSD together were given either verapamil or sertraline for 12 weeks. These medications are used to treat VM and CSD, though they are not approved for this purpose. Verapamil is believed to have stronger effects on symptoms of VM. Sertraline is believed to have stronger effects on symptoms of CSD. By comparing the responses of patients to these two medications, the researchers hoped to learn more about the key features of VM and CSD.

DETAILED DESCRIPTION:
Chronic dizziness and recurrent vertigo are frequent complaints in primary and specialty medical care settings. Two common causes of these symptoms are vestibular migraine (VM) and chronic subjective dizziness (CSD), which may be seen in up to 25% of patients examined in tertiary neurotology centers. However, VM and CSD are relatively new diagnoses that have not yet been validated. Furthermore, recent research found that they co-exist 30% of the time with overlap in several features. From a clinical standpoint, this makes it difficult to diagnose and treat them well. From a research standpoint, it confounds subject selection for mechanistic investigations.

The primary goal of this study was to dissect VM and CSD in order to identify the key features and clarify the diagnostic criteria of each condition. Subjects diagnosed with coexisting VM-CSD were treated with either verapamil or sertraline. It was hypothesized that a differential treatment response to these two pharmacologic probes would help to tease apart the unique clinical features of VM and CSD and identify risk factors that are shared or separate between the two conditions. It was hoped that the different mechanisms of action of the two study medications might also shed light on the physiologic underpinnings of VM and CSD.

This project was a 14-week, prospective, randomized, double-blind, parallel group, pharmacologic dissection (PD) trial. A 12-week treatment period followed 2 weeks of baseline observation. Patients charted daily headache and vestibular symptoms. VM and CSD symptoms and potential confounds such as anxiety and depression were measured at two week intervals. Data were analyzed for differential and shared treatment effects that align with or oppose current concepts of VM and CSD.

A PD trial uses response to one or more pharmaceutical probes (drugs) to study physiologic mechanisms of illness. A PD trial may provide data to separate overlapping manifestations of comorbid illnesses. This is useful for conditions that lack biomarkers. It also may provide data to identify characteristics of illnesses (symptoms, signs, cellular processes) that are associated with specific pharmacologic mechanisms.

ELIGIBILITY:
Inclusion criteria:

1. Neurotologic diagnoses of both vestibular migraine and chronic subjective dizziness
2. All other co-existing medical or psychiatric conditions are stable, and no greater than moderate severity
3. Able to complete study assessments in person and by phone
4. Able to travel to Mayo Clinic, Rochester, Minnesota for first and last study visits
5. Willing to avoid pregnancy during study (abstinence or acceptable birth control)

Exclusion criteria:

1. Presence of any other active neurotologic diagnoses
2. Medical or psychiatric conditions that would preclude or confound study drugs
3. Use of medications or supplements that would preclude or confound study drugs
4. Past treatment of headache or dizziness with a full trial of a calcium channel blocker or selective serotonin reuptake inhibitor
5. Allergy to verapamil or sertraline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
2-week Average Rating of Severity of Headache from the Daily Symptom Diaries | Week 0 to Week 12
  Daily ratings of headache will be evaluated at 2 week intervals for 12 weeks.
2-week Average Rating of Severity of Dizziness/Unsteadiness from the Daily Symptom Diaries | Week 0 to Week 12
  Daily ratings of dizziness/unsteadiness will be evaluated at 2 week intervals for 12 weeks.
2-week Average Rating of Sensitivity to Motion of Self from the Daily Symptom Diaries | Week 0 to Week 12
  Daily ratings of sensitivity to motion of self will be evaluated at 2 week intervals for 12 weeks.
2-week Average Rating of Sensitivity to Motion in the Environment from the Daily Symptom Diaries | Week 0 to Week 12
  Daily ratings of sensitivity to motion in the environment will be evaluated at 2 week intervals for 12 weeks.
2-week Average Rating of Difficulty of Performing Precision Visual Tasks from the Daily Symptom Diaries | Week 0 to Week 12
  Daily ratings of difficulty of performing precision visual tasks will be evaluated at 2 week intervals for 12 weeks.

SECONDARY OUTCOMES:
Mean Number of Acute Attacks Per Two Week Period | Week 0 to Week 12
  Acute attacks will be assessed every 2 weeks for 12 weeks.
Mean Score of Dizziness Handicap Inventory (DHI) | Week 0 to Week 12
  Dizziness related handicap will be assessed every 4 weeks for 12 weeks. The Dizziness Handicap Inventory (DHI) consists of 25 questions, with a total possible score ranging from 0 (no dizziness) to 50 (severe dizziness).
Mean Score of Migraine-Specific Quality of Life (MSQ) | Week 0 to Week 12
  Quality of life related to headache will be assessed at 4 week intervals for 12 weeks. The Migraine-Specific Quality of Life 2.1 (MSQ) consists of 14 items, with a total possible score ranging from 14 (affected none of the time) to 84 (affected all of the time).

OTHER OUTCOMES:
Mean score for Dizziness on the Sheehan Disability Scale/Migraine Disability Assessment Scale (SDS-MIDAS) | Week 0 to Week 12
  Dizziness symptoms will be assessed at 2 week intervals for 12 weeks. The Sheehan Disability Scale/Migraine Disability Assessment Scale (SDS-MIDAS) consists of 5 questions, with a total possible score ranging from 0 (no disability) to 72 (extremely disruptive).
Mean score for Headache on the Sheehan Disability Scale/Migraine Disability Assessment Scale (SDS-MIDAS) | Week 0 to Week 12
  Headache symptoms will be assessed at 2 week intervals for 12 weeks. The Sheehan Disability Scale/Migraine Disability Assessment Scale (SDS-MIDAS) consists of 5 questions, with a total possible score ranging from 0 (no disability) to 72 (extremely disruptive).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Staab, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Staab JP, Ruckenstein MJ. Expanding the differential diagnosis of chronic dizziness. Arch Otolaryngol Head Neck Surg. 2007 Feb;133(2):170-6. doi: 10.1001/archotol.133.2.170. PMID 17309987
- [Background] Ruckenstein MJ, Staab JP. Chronic subjective dizziness. Otolaryngol Clin North Am. 2009 Feb;42(1):71-7, ix. doi: 10.1016/j.otc.2008.09.011. PMID 19134491
- [Background] Eggers SD, Staab JP, Neff BA, Goulson AM, Carlson ML, Shepard NT. Investigation of the coherence of definite and probable vestibular migraine as distinct clinical entities. Otol Neurotol. 2011 Sep;32(7):1144-51. doi: 10.1097/MAO.0b013e31822a1c67. PMID 21799457